CLINICAL TRIAL: NCT02673853
Title: Assessment of Residual Paralysis in Patients Who Receive Mini-dose Atracurium During Supraglottic Airway Insertion
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/00055
Record Dates: First submitted 2016-01-04; First posted 2016-02-04 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Postoperative Complications
Keywords: Supraglottic airway; Mini-dose atracurium; Postoperative residual paralysis
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to establish the incidence of residual paralysis in patients following administration of a mini- dose of atracurium (less than ED95 i.e. <0.23mg/kg or <15 mg in most patients) during supraglottic airway insertion and correlate it with the duration of time from drug administration to arrival at PACU. The secondary aim is to compare the incidence of residual paralysis in patients who receive full doses of atracurium (per body weight) with those who receive mini-doses.

DETAILED DESCRIPTION:
Post-operative residual paralysis may be defined as the incomplete recovery of muscle function following intra-operative administration of neuromuscular blockers (NMBs). This condition is associated with many negative patient outcomes such as: increased risk of aspiration; upper airway obstruction; and delayed Post-Anaesthetic Care Unit (PACU) discharge, amongst others. Despite the increasing use of shorter acting agents, the prevalence of residual paralysis in the PACU remains high at 20-50%. NMBs are commonly used to facilitate endotracheal intubation and insertion of the supraglottic airway by obtunding airway reflexes. Given the increasing use of mini-dose NMBs without post-operative reversal in clinical practice, there is a need to evaluate the incidence of residual paralysis in the patient population who have received mini-dose atracurium during the supraglottic airway insertion.

ELIGIBILITY:
Inclusion Criteria:

* Adults above 21 years old
* Received either a mini-dose of atracurium or full dose of atracurium during the placement of the supraglottic airway
* Did not receive any neuromuscular reversal agent at any point of the operation.

Exclusion Criteria:

* Patients with underlying neuromuscular disease
* Patients who received pre-operative medication that may affect neuromuscular transmission
* Patients who required additional doses of neuromuscular blockade at any point of the operation

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be picked from all patients who are going surgery at National University Hospital (NUH) during the period of data collection, and who are receiving supraglottic airway for their procedure. They must fulfil the inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2016-02; Primary Completion 2018-03-08 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Number of patients with Post operative residual paralysis as measured by Train of Four (TOF) Ratio of < 0.9 | Through study completion, up to 4 months
  Measuring the extent of operative paralysis using established methods such as the train of four (TOF) with ratio of <0.9 indicating inadequate recovery, Double burst stimulation, acceleromyography, five second head lift and tongue depressor test. The relevant data about the patient's condition will be collected and filled up in the data collection form.

CONTACTS AND LOCATIONS:
Overall Officials: Lian Kah Ti, MBBS, MMed, Principal Investigator — National University Health System (NUHS)
Locations (1):
- National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Plaud B. Neuromuscular monitoring, residual blockade, and reversal: time for re-evaluation of our clinical practice. Can J Anaesth. 2013 Jul;60(7):634-40. doi: 10.1007/s12630-013-9952-4. Epub 2013 May 10. No abstract available. PMID 23661296
- [Background] Fortier LP, McKeen D, Turner K, de Medicis E, Warriner B, Jones PM, Chaput A, Pouliot JF, Galarneau A. The RECITE Study: A Canadian Prospective, Multicenter Study of the Incidence and Severity of Residual Neuromuscular Blockade. Anesth Analg. 2015 Aug;121(2):366-72. doi: 10.1213/ANE.0000000000000757. PMID 25902322
- [Background] Donati F. Residual paralysis: a real problem or did we invent a new disease? Can J Anaesth. 2013 Jul;60(7):714-29. doi: 10.1007/s12630-013-9932-8. Epub 2013 Apr 27. PMID 23625545